CLINICAL TRIAL: NCT06378086
Title: A Randomized, Controlled, Double-blinded, Within-subject (Split-face), Multicenter, Prospective Clinical Study to Compare the Level of Pain Using the Dermal Filler RHA® Redensity Formulated With Two Different Anesthetics in the Treatment of Perioral Rhytids
Brief Title: RHA® Redensity With New Anesthetic Agent Perioral Rhytids (PAS)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Teoxane SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TEO-PAS-2302
Record Dates: First submitted 2024-04-17; First posted 2024-04-22 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Pain; Aging
Keywords: Dermal filler; Perioral rhytids; Hyaluronic Acid; Anesthetic
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Split-face design
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- RHA® Redensity with new anesthetic agent (Experimental): Split-face injection of RHA® Redensity with new anesthetic agent in the perioral rhytids on one side of the mouth and RHA® Redensity with lidocaine in the perioral rhytids in the other side of the mouth.
  Up to 3 mL injected per side.
  Interventions: Device: RHA® Redensity with new anesthetic agent
- RHA® Redensity with lidocaine (Experimental): Split-face injection of RHA® Redensity with new anesthetic agent in the perioral rhytids on one side of the mouth and RHA® Redensity with lidocaine in the perioral rhytids in the other side of the mouth.
  Up to 3 mL injected per side.
  Interventions: Device: RHA® Redensity with lidocaine

INTERVENTIONS:
Device: RHA® Redensity with new anesthetic agent — A sterile, biodegradable, biocompatible, viscoelastic, clear, colorless, homogenized gel implant. It consists of cross-linked hyaluronic acid produced by fermentation of Streptococcus zooepidemicus, formulated to a concentration of 15 mg/g and 0.3% w/w of new anesthetic agent in a physiologic buffer.
  Arms: RHA® Redensity with new anesthetic agent
Device: RHA® Redensity with lidocaine — A sterile, biodegradable, biocompatible, viscoelastic, clear, colorless, homogenized gel implant. It consists of cross-linked hyaluronic acid produced by fermentation of Streptococcus zooepidemicus, formulated to a concentration of 15 mg/g and 0.3% w/w lidocaine in a physiologic buffer.
  Arms: RHA® Redensity with lidocaine

SUMMARY:
This is a randomized, controlled, double-blinded, within-subject (split-face), multicenter, prospective study to investigate whether RHA® Redensity with new anesthetic agent is non-inferior to RHA® Redensity with lidocaine in terms of injection site pain felt by the subject during injection.

At screening, the Principal Investigator (PI) evaluated subjects' perioral rhytid severity (using the Perioral Rhytid Severity Rating Scale; PR-SRS) to confirm eligibility and to establish a pre-treatment score for assessing aesthetic improvement.

At Visit 1, RHA® Redensity with new anesthetic agent was administered in a random sequence (first or second injection) and side of the mouth (left or right) and RHA® Redensity with lidocaine was administered to the other side. Study subjects and the PI injecting study devices were blinded.

Immediately after injection of an upper perioral quadrant, subjects rated the injection site pain experienced during injection using a 100 mm Visual Analog Scale (VAS). Injection site pain in each side of the mouth was also assessed at 15, 30, 45 and 60 minutes after injection of the upper quadrant.

Safety evaluation consisted of AE assessments, a 30-day CTR (Common Treatment Response) diary and a follow-up call performed by the study site at 72 hours after injection.

Subjects attended Visit 2 (30 days post-injection) where effectiveness and safety assessments were conducted.

Subjects who presented with an unresolved clinically significant device related AE at Visit 2 received a optional follow-up phone call no later than 30 days after Visit 2.

If the clinically significant AE remained unresolved, the Investigator requested that the subject attended the optional in-clinic follow-up visit (i.e., Visit 3) within 5 working days. Follow-up of the clinically significant AE continued until the AE was resolved or the TI determines that additional follow-up was not necessary.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatient, male or female of any race, 22 years of age or older. Female subjects of childbearing potential must have a negative UPT at Visit 1 and practice a reliable method of contraception throughout the study.
2. Perioral rhytids of the same PR-SRS grade on the left and right sides of the mouth.
3. Able to follow study instructions and complete all required visits.
4. Sign the IRB-approved ICF, Photographic Release Form, the Authorization for Use and release of Health and Research Study Information (HIPAA) form, and if applicable the California Experimental Research Subject's Bill of Rights prior to any study-related procedures being performed.

Exclusion Criteria:

1. Female subjects who are pregnant, breast-feeding, or of childbearing potential and not practicing reliable birth control.
2. Known hypersensitivity or previous allergic reaction to any component of the study devices.
3. Known sensitivity to local anesthetics of the amide type, history of multiple severe allergies, or history of anaphylactic shock.
4. Clinically significant active skin disease or infection in the perioral area within 6 months prior to study entry (TI discretion).
5. History of active chronic debilitating systemic disease that, in the opinion of the investigator, would make the subject a poor candidate in the study.
6. Malignancy (excluding non-melanoma skin cancer) within the past 5 years.
7. History or presence of condition or feature that may confound the interpretation of the results in the perioral region, for example, tattoo, significant facial hair, acne scaring, prior surgery in the area, potential for active disease or infection flare up such as herpes simplex.
8. History of skin cancer in the treatment area.
9. Elective, clinically significant facial procedures that may confound the interpretation of the results in the perioral region (TI discretion), prior to study enrollment.
10. Clinically active disease or infection in the perioral area or mouth (e.g., dental abscess).
11. Clinically significant alcohol or drug abuse, or history of poor cooperation or unreliability.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-11 (Actual); Primary Completion 2025-02-26 (Actual); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Non-inferiority of RHA® Redensity with new anesthetic agent versus RHA® Redensity with lidocaine in terms of reducing pain during device injection into the upper perioral rhytids. | Visit 1 - During Injection
  Injection pain during injection was measured on the 100 mm Visual Analog Scale (VAS), as assessed by subjects immediately after injection of each upper perioral quadrant.
  VAS is a 100 mm Visual Analog Scale with 0 meaning no pain and 100 meaning intolerable pain

SECONDARY OUTCOMES:
Difference between RHA® Redensity with new anesthetic agent versus RHA® Redensity with lidocaine in term of reducing pain at 15, 30, 45 and 60 minutes post-injection in each side of the mouth. | Visit 1 - 15, 30, 45 and 60 minutes post-injection
  Injection pain was measured on the 100 mm Visual Analog Scale (VAS), as assessed by subjects in each side of the mouth.
  VAS is a 100 mm Visual Analog Scale with 0 meaning no pain and 100 meaning intolerable pain

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - United States, Birmingham, Alabama
  - United States, New York, New York, New York
- Puerto Rico, San Juan, Puerto Rico